| Cover page |
|---|
| Title: Individual Follow-up after Rectal Cancer - Focus on the Needs of the Patient (FURCA) |
| [NCT-number not assigned yet] |
| Date: 06 January 2016 |

## Informed consent for participation in a health science research project.

The research project title: "Individualized follow-up after rectal cancer - focus on the needs of the patients"

## **Declaration from participant in the survey:**

I have received written and oral information and I have sufficient knowledge about the purpose, method, advantages and disadvantages in order to accept participation.

I am aware that it is voluntary to participate and that I at any time can withdraw my consent without compromising the rights to any current or future treatment.

I agree to participate in the research study and have received a copy of this consent sheet as well as a copy of the written information on the study for my own use.

| Name of the participant: |
|---|
| Determined allowed ways |
| Date and signature: |
| Do you want to be informed about the results of the study and any consequences for you?: |
| Yes (set x) No (set x) |
| Declaration from the person providing information: I declare that the participant has received oral and written information about the study. |
| In my belief, sufficient information has been provided for a decision to participate in the investigation. |
| The name of the person who provided information: |
| Date and signature: |
| Project Identification: FURCA 06.01.2016 |